CLINICAL TRIAL: NCT06520917
Title: Evaluating the Accuracy and Safety of a Locator-Positioner Guide Device to Assist in Temporomandibular Joint Arthroscopy
Brief Title: Novel Locator-Positioner Device for Temporomandibular Joint Arthroscopy
Acronym: TMJ-LOPO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: SMC-4657-17; 93765 (Other Grant/Funding Number: Sheba Medical Center)
Record Dates: First submitted 2024-07-21; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2018-04

CONDITIONS: Temporomandibular Joint Disc Displacement; Temporomandibular Joint Disorders; Temporomandibular Joint Dysfunction Syndrome
Keywords: Arthroscopy; Arthroscopic surgery; Temporomandibular joint closed lock; Temporomandibular joint
MeSH Terms: conditions — Temporomandibular Joint Disorders; Temporomandibular Joint Dysfunction Syndrome

STUDY DESIGN:
Intervention Model Description: Patients that were included in the study underwent temporomandibular joint arthroscopy using the Locator-Positioner Device, as opposed to the usual/classic procedure of temporomandibular joint arthroscopy without the aid of the Locator-Positioner Device
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Performing temporomandibular joint arthroscopy with the aid of the Locator-Positioner (LOPO) Device (Experimental): The patients underwent the arthroscopic procedure of the temporomandibular joint with the guidance of the Locator-Positioner Device
  Interventions: Device: Locator-Positioner (LOPO) Guide Device

INTERVENTIONS:
Device: Locator-Positioner (LOPO) Guide Device — Patients underwent temporomandibular joint arthroscopy with the aid of the LOPO guide device

SUMMARY:
The goal of this clinical trial is to evaluate a guide device (locator-positioner LOPO guide device) that is intended to aid the surgeon in temporomandibular joint (TMJ) arthroscopy. The aim of the device is to help the surgeon introduce the arthroscope and working cannula into the TMJ space. The trial evaluates the accuracy and safety of the device.

The main questions it aims to answer are:

* Does the LOPO guide device increase the accuracy of inserting the arthroscope and working cannula into the temporomandibular joint?
* Does the number of attempts to correctly place the working cannula relative to the arthroscope decrease?
* Does the overall time of surgery decrease when using the LOPO device?
* Does the device pose new surgical risks to temporomandibular joint arthroscopy?

The LOPO device was tried on anatomical models and proved to be very accurate. The present study recruits up to 10 patients to participate in this experiment. IRB approval and Ministry of Health approval have been given for conducting the clinical trial in 10 patients.

Participants will:

* Have a diagnosis of temporomandibular closed lock based on clinical and imaging findings.
* Undergo temporomandibular joint arthroscopy with the aid of the LOPO device.
* Visit the clinic for routine follow-up visits after roughly 1 week, 3 weeks, 2 months, and 6 months postoperatively, and at each visit be evaluated for maximal mouth opening and severity of pain on a 1-10 VAS.

DETAILED DESCRIPTION:
Temporomandibular joint arthroscopy allows for direct visualization and access to the joint, enabling surgeons the ability to diagnose and perform a wide range of procedures. Arthroscopic surgery mandates the insertion of at least two portals into the joint cavity. The first is the arthroscope and is usually made through a lateral approach into the posterior recess of the superior joint space. Generally this is an easy puncture as the glenoid fossa is easily palpated and the target point is just deep to the skin and joint capsule. The second puncture is intended to incorporate the working cannula, through which instruments are introduced into the joint cavity, and is generally targeted to the anterior recess of the superior joint space. For the second or working cannula to be readily visualized by the arthroscope and functional, skin puncture site, angulation of insertion, and insertion depth must be accurate and precise. The site and technique of the second puncture are dictated by the anatomy and volume of the anterior recess of the superior joint space which has great variability between individuals and joint conditions. The target point is the juncture between the anterior aspect of the anterior slope of the articular eminence and the continuation of the zygoma, which is generally not palpable. To overcome this difficulty, the triangulation technique was adapted for the temporomandibular joint by pioneer arthroscopists such as K Murakami and J P McCain. The rationale behind using it was to facilitate easier and more predictable entry of the second portal to avoid unnecessary scuffing or damaging of the joint surfaces. It enables a repeatable, safe, and strategic insertion and placement for the second cannula that provides access to different areas in the joint while being fully visualized by the arthroscope.

Adherence to the triangulation principles is essential for achieving a successful placement of the second or working cannula. However, it takes a considerable amount of time to become proficient in this technique. Furthermore, maintaining the optimal spatial alignment of the working cannula with the arthroscope throughout the surgery necessitates additional practice, experience, and synchronized collaboration between the surgeon and assistant.

The main author developed a Locator-Positioner (LOPO) guide device to assist the surgeon in inserting the working cannula and in maintaining its' three-dimensional position relative to the arthroscope throughout surgery, while permitting movement of both portals. The desired benefit was to achieve an easy and accurate method to insert and position the working cannula and help minimize intra-articular scuffing and surgical risks. The purpose of the present study was to examine the accuracy, safety, and efficiency of the LOPO guide device.

The guide device consists of two arms of equal length, each being a double parallelogram. A connector holds both arms and permits movement by changing the angle between them. One arm is intended to hold the arthroscope while the other is intended for the insertion of the working cannula. After the arthroscope is introduced into the joint cavity, the guide device is mounted on the base of the arthroscope via one arm. The other arm receives the working cannula, and owing to the double parallelogram design, it directs it to the ideal puncture site and insertion vector and depth into the joint cavity, where it has to meet the tip of the arthroscope. This results in immediate visualization of the working cannula by the arthroscope and maintains optimal spatial positions between the two portals. The connector between the two arms of the device enables changing the angle between them while maintaining the relative position of the tip of the cannula to the tip of the arthroscope. The connector can also be locked thus fixating the angle between the two arms.

During surgery, the surgeon holds the LOPO device with the two cannulas mounted on it with one hand, while the other hand is free to perform surgical instrumentation through the working cannula. All this is performed while the ideal position of the working cannula relative to the arthroscope is maintained due to the double parallelogram design. The guide device can be mounted and dismounted at any time during the operation without the need to remove the cannulas from the joint. It is a Patent No. US 11,517,348 B2.

Approval for conducting an experiment with human subjects using the LOPO device was granted by the Institutional Review Board (IRB approval 4657-17-SMC) and the National Ministry of Health (MOH_2018-08-27_003619). The clinical trial was registered before enrolment of patients.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with closed lock of the temporomandibular joint (Wilkes stage III internal derangement) based on clinical examination and MRI findings.
* Subjects accepting to participate in the study and undergoing the arthroscopic procedure with the aid of the LOPO device.
* Subjects that are adults (> 18 years), not pregnant, and of sound judgement.

Exclusion Criteria:

* Diagnosis of other temporomandibular joint disorders.
* Minor patients under 18 years.
* Pregnant patients.
* Subjects lacking sound judgement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-08-31 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2020-01-18 (Actual)

PRIMARY OUTCOMES:
Number of attempts made to successfully insert the working cannula into the joint space | This outcome is reported during the surgical procedure, as the number of attempts is counted by a resident in the operating room
  After puncturing the skin and advancing to the joint, any partial or complete withdrawal of the cannula followed by a change of vector or depth was considered an additional attempt. Confirmation of successful insertion was based on visualizing the working cannula by the arthroscope (i.e. observing the working cannula on the monitor).
The duration of time between the arthroscope's insertion into the joint cavity and the initial appearance of the working cannula on the monitor. | This outcome is reported during the surgical procedure, as the time is measured by a resident in the operating room
  The time that elapsed from the point when the arthroscope was inserted in the joint space and the point when the working cannula was seen on the monitor.

CONTACTS AND LOCATIONS:
Overall Officials: Waseem Abboud, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: Yes
Data of the 10 subjects participating in the research will be sent via email upon request to other researchers. Data that can be shared (for each participant):
  * Age
  * Gender
  * Duration of closed lock of the temporomandibular joint
  * Maximal mouth opening before arthroscopy
  * Maximal mouth opening after arthroscopy
  * Number of attempts made to correctly position the working cannula relative to the arthroscope
  * The time duration between the insertion of the arthroscope and visualization of the working cannula by it
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data is available. It will remain available for 1 year after publishing the study in an international medical journal.
Access Criteria: A researcher that identifies with an ORCID ID and an email of an academic institution identified by the email's suffix.

REFERENCES:
- [Background] Abboud WA. Novel guide device for temporomandibular joint arthroscopy. Int J Oral Maxillofac Surg. 2020 Sep;49(9):1217-1219. doi: 10.1016/j.ijom.2020.02.013. Epub 2020 Mar 11. PMID 32171619
- [Background] Monje Gil F, Hernandez Vila C, Moyano Cuevas JL, Lyra M, Pagador JB, Sanchez Margallo FM. Validation of a simulator for temporomandibular joint arthroscopy. Int J Oral Maxillofac Surg. 2016 Jul;45(7):836-41. doi: 10.1016/j.ijom.2016.01.010. Epub 2016 Feb 3. PMID 26850940
- [Background] Verde L, Munoz-Guerra MF, Rodriguez-Campo FJ, Escorial V. Temporomandibular Joint: Approach to the Intermediate Space by Triangulation With Transillumination Reference. J Oral Maxillofac Surg. 2023 Jun;81(6):684-688. doi: 10.1016/j.joms.2023.02.008. Epub 2023 Mar 6. PMID 36893793
- [Background] Peserico-DalFarra P, Gagliardi-Lugo AF. Training simulation for oral and maxillofacial surgeons based on the techniques of arthroscopy in the temporomandibular joint. Br J Oral Maxillofac Surg. 2019 Nov;57(9):929-931. doi: 10.1016/j.bjoms.2019.08.003. Epub 2019 Aug 22. PMID 31445774
- [Background] Slavin AB. Comments on "single-cannula technique for operative arthroscopy using holmium:YAG laser". J Oral Maxillofac Surg. 2012 May;70(5):1014; author reply 1014. doi: 10.1016/j.joms.2012.02.011. No abstract available. PMID 22538020
- [Background] McCain JP, Hossameldin RH. Advanced arthroscopy of the temporomandibular joint. Atlas Oral Maxillofac Surg Clin North Am. 2011 Sep;19(2):145-67. doi: 10.1016/j.cxom.2011.06.001. No abstract available. PMID 21878249
- [Derived] Abboud W, Reiter S, Friedman-Rubin P, Shamir D, Peleg O. Guide device to assist in performing arthroscopic surgery of the temporomandibular joint-a preliminary study. J Oral Facial Pain Headache. 2025 Mar;39(1):128-133. doi: 10.22514/jofph.2025.012. Epub 2025 Mar 12. PMID 40129430

DOCUMENTS (1):
  • Study Protocol (2018-03-09): https://cdn.clinicaltrials.gov/large-docs/17/NCT06520917/Prot_000.pdf